CLINICAL TRIAL: NCT00249470
Title: The Therapeutic Workplace Initiation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WIRB 2162; R01DA012564 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Cocaine-Related Disorders; Opioid-Related Disorders; Heroin Dependence; Substance Abuse, Intravenous
Keywords: HIV; HIV risk behaviors; Heroin; Cocaine; Methadone; Opioid Dependence; Cocaine Abuse; Contingency management; alcohol & drug use; sexual risk behaviors
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Heroin Dependence; Substance Abuse, Intravenous; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abstinence & Work (Experimental): Participants in the Abstinence & Work group were invited to attend the workplace throughout a 26-week intervention period, but were required to provide urine samples that indicated recent cocaine abstinence to gain access to the workplace and to maintain the maximum base pay of $8.00 per hour.
  Interventions: Behavioral: Abstinence & Work
- Work Only (Other): Work Only participants were invited to attend the workplace throughout a 26-week intervention period. Participants in this group continued to provide mandatory urine samples and could earn base and performance pay. Work Only participants could work and earn base and performance pay independent of urinalysis results.
  Interventions: Behavioral: Work Only

INTERVENTIONS:
Behavioral: Abstinence & Work — Participants in the Abstinence & Work group were invited to attend the workplace throughout a 26-week intervention period, but were required to provide urine samples that indicated recent cocaine abstinence to gain access to the workplace and to maintain the maximum base pay of $8.00 per hour.
  Arms: Abstinence & Work
Behavioral: Work Only — Work Only participants were invited to attend the workplace throughout a 26-week intervention period. Participants in this group continued to provide mandatory urine samples and could earn base and performance pay. Work Only participants could work and earn base and performance pay independent of urinalysis results.
  Arms: Work Only

SUMMARY:
The primary purpose of the study is to determine if the central feature of the Therapeutic Workplace, the abstinence reinforcement contingency, is critical to initiate cocaine abstinence in injection drug using methadone patients who use cocaine consistently during methadone treatment. All subjects initially will be invited to attend the Therapeutic Workplace for an initial period, but abstinence will not be required to work during that time. During this initial period, vouchers will be contingent only on workplace attendance and performance on the training programs. Subjects (n=70) who attend the workplace consistently during the first 4 weeks of treatment, but who continue to use cocaine will be randomly assigned to a Work Only or an Abstinence Plus Work group. Subjects in the Work Only group will continue to be able to work independent of their urinalysis results. However, subjects in the Abstinence Plus Work group will be required to provide urine samples that show evidence of recent cocaine abstinence. Subjects in both groups will be invited to stay in the workplace for 6 months. We expect the subjects in the Abstinence and Work group will achieve higher rates of abstinence than the subjects in the Work Only group. This result would show that the abstinence reinforcement contingency (i.e., the requirement to provide cocaine-free urine samples to work and earn vouchers) is important in the initiation of abstinence in the study population.

DETAILED DESCRIPTION:
Methods Setting and Materials This study was conducted at the Center for Learning and Health, a treatment-research unit at the Johns Hopkins Bayview Medical Center, Baltimore, MD. The therapeutic workplace included a workplace sign-in station and urinalysis laboratory, and three workrooms (and associated staff space) where training occurred. When participants arrived at the workplace each day, they reported to the workplace sign-in station located at the entrance to the urinalysis laboratory. Staff sat on the laboratory side of the entrance at the workplace sign-in station desk, which was equipped with a Dell personal computer and electronic barcode reader (Unitech® Barcode Slot Reader model # MS140I-2, St Louis, MO).

Urine and breath samples were collected and tested in the urinalysis laboratory. Breath samples were tested for alcohol with the AlcoSensor III (Intoximeter, St. Louis, MO). Females provided urine samples directly into Commode Specimen Containers (Catalog #00077, Sage Products, Inc., Crystal Lake, IL) that were placed directly on the toilet. The urine samples were then temperature tested and transferred to storage cups. Males provided samples directly into paper cups, which were then temperature tested and transferred to storage cups. All urine samples were temperature tested using an F-1500 Electronic Thermometer (Sherwood Medical, St. Louis, MO). The urinalysis laboratory contained an Abbott AxSYM® immunoassay system for urine testing. The AxSYM® employs fluorescent polarization immunoassay (FPIA) technology (Abbott Laboratories, Abbott Park, IL).

Participants received the therapeutic workplace training programs in three workrooms (a total of 161 m2) that contained a total of 47 individual three-sided workstations (155 cm tall x 64 cm deep x 126 cm wide). Each workstation was equipped with a desktop (60 cm deep x 121 cm wide); a height adjustable chair with arms; a Dell personal computer, keyboard and mouse. Keyboards were covered with removable plastic covers (Protect Keyboard Cover, West Bountiful, UT) that were painted black that so that the letters on the keys could not be read while typing. Each participant was given a water bottle, headphones for listening to music CDs during training on the personal computer, a cooler for storing lunch, and picture frames to personalize the workstation.

The three workrooms opened into a central area (31 m2) where the workroom assistants sat to monitor the activities of participants in the workrooms. Participants had to pass through the central staff area to enter and leave the workrooms. The central area was equipped with three desks, each with a personal computer. Each desk also was equipped with a Unitech® electronic barcode slot reader.

All of the participant and staff computers were interconnected through a high-speed (T1) line to central Dell PowerEdge servers. All of the typing, keypad and data entry training programs; monitoring of the work time and earnings; and the voucher system were controlled by a custom web-based therapeutic workplace software application program that resided on one of the PowerEdge servers (Silverman et al., 2005).

Recruitment and Participant Selection The Western Institutional Review Board approved this study. Participants were enrolled in this study from April 2003 to November 2003. To recruit participants, flyers and letters were distributed to 11 Baltimore City methadone programs inviting unemployed adults in methadone treatment to apply to enroll in a study that provided job skills training and monetary vouchers. Research staff also visited the methadone treatment programs to describe the study to methadone treatment staff (e.g., counselors).

Interested individuals who approached or called research staff first completed an anonymous brief screening interview in which they were asked 8 questions designed to determine quickly if they might be eligible for the study. Some of the questions were added to conceal the eligibility requirements. The interview asked the individuals' age, marital status, employment status, drugs and routes of administration used in the past 30 days, what type of drug abuse treatment they currently receive, whether they receive welfare benefits, how much they earned through employment in the past 30 days, and whether they have any of several medical conditions (e.g., asthma, HIV). Brief screening interviews were conducted over the phone, in person at the methadone treatment programs, or in person at the Center for Learning and Health. Applicants were invited to participate in a full screening interview if they reported that they were 18 years or older, were unemployed, injected heroin or cocaine, used cocaine or crack in the past 30 days, and if they were currently enrolled in methadone maintenance treatment in Baltimore City.

Full screening interview. At the beginning of the full screening interview, participants were invited to sign the initial screening consent form. Participants were required to pass a written quiz about the details of the consent form to participate. Participants were also required to read a paragraph of the consent form aloud and to read at least 80% of the words correctly to continue in the full screening interview.

Baseline period. Eligible participants were invited to attend the workplace for 4 hours every weekday for 8 weeks. Mandatory urine samples were collected prior to work every Monday, Wednesday and Friday. All samples were tested for cocaine and opiates. During the first 4 weeks, participants could attend the workplace independent of their urinalysis results and earn a base pay of $8.00 per hour plus pay for performance on training programs. To encourage brief breaks, participants could earn 5 minutes of paid break for every 55 minutes worked. Pay was earned in vouchers exchangeable for goods and services. At the end of baseline, participants who attended the workplace at least 50% of the workdays, provided at least two cocaine-positive urine samples, and were still enrolled in methadone treatment were invited to participate in the main randomized controlled portion of the study. Other participants could continue to work for 4 additional weeks, but were required to provide urine samples that indicated recent abstinence from opiates and cocaine to work.

Experimental Design and Groups Stratification and random assignment. Participants enrolled in the main study (N = 56) were randomly assigned to the Work Only (n = 28) or Abstinence & Work (n = 28) group. Immediately prior to actual assignment, a study coordinator, who did not have direct contact with participants, randomized participants using a computer program and a stratification procedure (similar to Silverman et al., 2004) based on a) whether 75% or more of the participant's baseline urine samples tested positive for cocaine (Y/N), and b) whether 100% of the participant's baseline urine samples tested positive for cocaine (Y/N).

Study groups. Both groups were invited to attend the workplace throughout a 26-week intervention period. Participants in both groups continued to provide mandatory urine samples and could earn base and performance pay. Both groups also received the same feedback as to the results of the urinalysis testing. The two groups differed only in that participants in the Abstinence & Work group were required to provide urine samples that indicated recent cocaine abstinence (i.e., decreased urinary benzoylecgonine concentration of 20% per day from the last sample provided or benzoylecgonine concentration at or below 300 ng/mL; adapted from procedures developed by Preston, Schuster, Silverman & Cone, 1997) to gain access to the workplace and to maintain the maximum base pay of $8.00 per hour. If the participant ever provided a urine sample that did not meet the criteria for recent cocaine abstinence or if the participant failed to provide a scheduled sample, the participant was not allowed to work that day and the participant's base pay was decreased to $1.00 per hour. In addition, the participant was required to provide a urine sample every workday until the participant provided a sample that met the abstinence requirement. After a participant's base pay was reset, it increased by $1.00 per hour to a maximum of $8.00 per hour for every day that the participant met the cocaine abstinence requirement and worked at least 5 minutes. The voucher system and the schedule of escalating reinforcement for sustained abstinence and workplace attendance was adapted from a system developed by Higgins et al., 1991.

General Workplace Procedures Urine collection, testing and feedback. After signing into the workplace on mandatory urine days (typically Monday, Wednesday and Friday of each week), participants were required to provide a urine and breath sample under observation by a same-gender research staff member. Urine collection was performed using well-developed and elaborate urine-collection procedures designed to ensure the collection of valid urine samples. Urine samples were tested for cocaine and opiates.

For participants who had to provide evidence of recent cocaine abstinence to enter the workroom, immediately after the participant provided the urine sample, the sample was tested and the results (i.e., the quantitative value in ng/mL for benzoylecgonine and the dichotomous result of negative or positive for opiates) were entered into the therapeutic workplace software. The software automatically determined whether or not the sample met the cocaine abstinence criterion for that day, displayed a message reporting the result of that determination, and printed a feedback graph to be given to the participant. The feedback graph showed on a log scale the benzoylecgonine concentrations of all samples provided by the participant over consecutive calendar days, along with a line indicating the criterion for cocaine abstinence for each of the days. In addition, a text box was printed to the side of the graph that indicated the results for the current day including the benzoylecgonine concentration, whether the sample tested negative or positive for opiates, and if the participant was granted access to the workplace. If the sample met the cocaine abstinence requirement, the sign-in station assistant gave the participant his or her bar-coded picture ID card to bring to the workroom assistant to gain entrance to the participant's workroom.

During conditions in which there were no contingencies on cocaine abstinence to gain access to the workplace (i.e., during the baseline period and during the intervention period for the Work Only participants), immediately after a participant provided a urine sample and before the sample was tested, the sign-in station assistant handed the participant his or her bar-coded picture ID card to bring to the workroom assistant to gain entrance to the participant's workroom. Later that day, the participant's sample was tested, the results were entered into the therapeutic workplace software, and a feedback graph (identical to the one described above) was printed and delivered to the participant.

ELIGIBILITY:
Baseline inclusion criteria:

* are at least 18 years of age
* are enrolled in methadone maintenance treatment in Baltimore
* provide a cocaine-positive urine sample at time of initial screening
* self-report cocaine use through intravenous route
* have visible evidence of intravenous drug use (i.e., track marks).

Baseline exclusion criteria:

* report current suicidal ideation
* if the individual reports hallucinations
* have physical limitations (e.g., broken fingers) that prevent the subject from typing.
* Applicants reporting hallucinations are excluded because this is a characteristic of a psychiatric disorder that is likely to result in behaviors that could disrupt the workplace or functioning or limit their ability to provide informed consent.

Main study inclusion criteria:

* have attended the workplace regularly during 4-week baseline periods
* are still in methadone maintenance treatment at the end of the 4-week baseline period
* have provided at least two urine samples that test positive for cocaine during the baseline period
* Individuals who are excluded from the main study will be allowed to complete their 8-week training program in the Therapeutic Workplace. They may also be invited to participate in other studies ongoing at the Center for Learning and Health where this research takes place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2003-04; Primary Completion 2004-05 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silverman K, Wong CJ, Needham M, Diemer KN, Knealing T, Crone-Todd D, Fingerhood M, Nuzzo P, Kolodner K. A randomized trial of employment-based reinforcement of cocaine abstinence in injection drug users. J Appl Behav Anal. 2007 Fall;40(3):387-410. doi: 10.1901/jaba.2007.40-387. PMID 17970256

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 completed the induction period and were randomly assigned to the two study groups.
Period: Overall Study
Arm/Group | Abstinence & Work | Work Only
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abstinence & Work | Work Only | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (6.5) | 47.5 (5.8) | 45.7 (6.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Abstinence
Description: Percentage of Monday, Wednesday, Friday urine samples that are negative for cocaine
Time Frame: 6 months
Measure: Mean (Full Range); unit: percentage of cocaine negative
Arm/Group | Abstinence & Work | Work Only
Number analyzed (Participants) | 28 | 28
percentage of cocaine negative | 29 [0 to 99] | 10 [0 to 64]
Statistical Analysis 1: Comparison: Abstinence & Work vs Work Only; Test type: Superiority or Other; p = .004, General Estimating Equation (GEE); Odds Ratio (OR) = 5.80, 95% CI 2-sided [2.03 to 16.56]

2. Secondary Outcome: Percent Opiate Negative
Description: (total number of opiate-negative urine samples divided by the total number of urine samples provided)*100
Time Frame: every month for 6 months
Population: intent to treat
Measure: Mean (Full Range); unit: percentage of opiate negative
Arm/Group | Abstinence & Work | Work Only
Number analyzed (Participants) | 28 | 28
percentage of opiate negative | 55.4 [0 to 100] | 62.5 [0 to 100]
Statistical Analysis 1: Comparison: Abstinence & Work vs Work Only; Test type: Superiority; p = 0.82, General Estimating Equation (GEE); Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.40 to 2.08]

3. Secondary Outcome: HIV Risk Behaviors
Description: Report no injection drug use or crack cocaine use.
Time Frame: every month for 6 months
Population: The data represent the mean percentage of participants that reported no injection drug use or crack cocaine use. Missing assessments were considered positive (i.e., injection drug or crack cocaine use).
Measure: Mean (Full Range); unit: percentage of participants
Arm/Group | Abstinence & Work | Work Only
Number analyzed (Participants) | 28 | 28
percentage of participants | 28.0 [0 to 78] | 16.1 [0 to 67]
Statistical Analysis 1: Comparison: Abstinence & Work vs Work Only; Test type: Superiority; p = 0.04, General Estimating Equation (GEE); Odds Ratio (OR) = 3.37, 95% CI 2-sided [1.21 to 9.37]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Abstinence & Work | Work Only
Serious Adverse Events (participants affected / at risk) | 4/28 | 2/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abstinence & Work (N=28) | Work Only (N=28)
Death from heart attack (Cardiac disorders) | 1 (1) | 0 (0) — Death occurred about 5 months after leaving the study.
Hospitalization for congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) — Not related
Hospitalization for abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not related
Hospitalization for general medical treatment (General disorders) | 1 (1) | 1 (1) — Not related
Hospitalization for inpatient surgery (General disorders) | 1 (1) | 0 (0) — Not related
Hospitalization for infection (Infections and infestations) | 0 (0) | 1 (1) — Not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No